CLINICAL TRIAL: NCT04895449
Title: A Multi-center Phase Ib Trial to Assess the Safety, Tolerability and Immunogenicity of the Candidate Vaccine MVA-SARS-2-ST in Adults
Brief Title: Safety, Tolerability and Immunogenicity of the Candidate Vaccine MVA-SARS-2-ST Against COVID-19
Acronym: MVA-SARS2-ST
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: German Center for Infection Research (Other); Philipps University Marburg (Other); Ludwig-Maximilians - University of Munich (Other); IDT Biologika (Unknown); Clinical Trial Center North (CTC North GmbH & Co. KG) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UKE-SARS-CoV-2-ST
Record Dates: First submitted 2021-04-24; First posted 2021-05-20 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Covid19
Keywords: MVA; SARS-CoV-2; vaccine; booster vaccination
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- ≥ 1 x 10E7 IU (low dose) in seronegative subjects (Experimental): ≥ 1 x 10E7 IU MVA-SARS-2-ST Intervention: Biological: MVA-SARS-2-ST vaccinations (days 0 & 28) in seronegative subjects
  Interventions: Biological: MVA-SARS-2-ST
- ≥ 5 x 10E7 IU (middle dose) in seronegative subjects (Experimental): ≥ 5 x 10E7 IU MVA-SARS-2-ST Intervention: Biological: MVA-SARS-2-ST vaccinations (days 0 & 28) in seronegative subjects
  Interventions: Biological: MVA-SARS-2-ST
- ≥ 1 x 10E8 IU (high dose)in seronegative subjects (Experimental): ≥ 1 x 10E8 IU MVA-SARS-2-ST Intervention: Biological: MVA-SARS-2-ST vaccinations (days 0 & 28) in seronegative subjects
  Interventions: Biological: MVA-SARS-2-ST
- ≥ 1 x 10E7 IU (low dose) (Experimental): ≥ 1 x 10E7 IU MVA-SARS-2-ST Intervention: Biological: Single MVA-SARS-2-ST vaccination in mRNA vaccinated subjects
  Interventions: Biological: MVA-SARS-2-ST
- ≥ 5 x 10E7 IU (middle dose) (Experimental): ≥ 5 x 10E7 IU MVA-SARS-2-ST Intervention: Biological: Single MVA-SARS-2-ST vaccination in mRNA vaccinated subjects
  Interventions: Biological: MVA-SARS-2-ST
- ≥ 1 x 10E8 IU (high dose) (Experimental): ≥ 1 x 10E8 IU MVA-SARS-2-ST Intervention: Biological: Single MVA-SARS-2-ST vaccination in mRNA vaccinated subjects
  Interventions: Biological: MVA-SARS-2-ST

INTERVENTIONS:
Biological: MVA-SARS-2-ST — i.m. vaccine administration

SUMMARY:
Multi-center phase Ib study to evaluate the Modified Vaccinia Virus Ankara (MVA) vaccine against SARS-CoV-2 in seronegative (Part A) and previously SARS-CoV-2-vaccinated individuals (Part B).

DETAILED DESCRIPTION:
The vaccine contains a Modified Vaccinia Virus Ankara (MVA) vector expressing a stabilized SARS-CoV-2 spike protein (S).

This will be a phase Ib multi-center study in approximately 60 adults aged 18-64 years.

Part A (N=24 seronegative subjects). Each participant will receive two single injections, 28 days apart.

* low dose ≥ 1 x 10e7 IU (N=8)
* middle dose ≥ 5 x 10e7 IU (N=8)
* high dose ≥ 1 x 10e8 IU (N=8)

Part B (N=36 previously mRNA vaccinated subjects). Each participant will receive a single injection.

* low dose ≥ 1 x 10e7 IU (N=12)
* middle dose ≥ 5 x 10e7 IU (N=12)
* high dose ≥ 1 x 10e8 IU (N=12)

All participants will be followed up for safety until D168.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Healthy male and female adults aged 18 - 64 at time of informed consent.
3. Body mass index 18.5 - 32.0 kg/m2 and weight > 50 kg at screening.
4. Female participants: non-pregnant, non-lactating with negative pregnancy test.
5. Females who agree to comply with the applicable contraceptive requirements of the protocol.
6. ≥ 6 months fully vaccinated with a (conditionally)licensed mRNA vaccine against COVID-19 (Part B only)

Exclusion Criteria:

1. Receipt of any vaccine from 4 weeks prior to each trial vaccination (8 weeks for live vaccines) to 6 weeks after each trial vaccination.
2. Previous rMVA immunization.
3. Previous immunization with investigational vaccine against COVID-19.
4. Previous immunization with EUA/conditionally licensed vaccine against COVID-19 (not applicable to Part B).
5. Evidence of active SARS-CoV-2 infection
6. Known allergy to the components of the MVA-SARS-2-ST vaccine product or history of life-threatening reactions to vaccine containing the same substances.
7. Known history of anaphylaxis to vaccination or any allergy likely to be exacerbated by any component of the trial vaccines.
8. Evidence in the participant's medical history or in the medical examination that might influence either the safety of the participant or the absorption, distribution, metabolism or excretion of the investigational product.
9. Clinically relevant findings in ECG or significant thromboembolic events in medical history.
10. Any confirmed or suspected immunosuppressive or immunodeficient condition, cytotoxic therapy in the previous 5 years, and/or uncontrolled diabetes (HbA1c ≥ 7.0).
11. Any known chronic or active neurologic disorder, including seizures and epilepsy, excluding a single febrile seizure as a child.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2021-07-16 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2022-11-08 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Experiencing Solicited Local or Systemic Reactogenicity as Defined by the Study Protocol | during the entire study (up to 6 months)
  Safety and reactogenicity will be assessed by observation, questionaire and diary. Occurence of Serious Adverse Events (SAE) will be collected throughout the entire study duration.

SECONDARY OUTCOMES:
Number of participants who seroconverted | during the entire study (up to 6 months)
  Magnitude of SARS-CoV-2-S specific antibody responses will be measured by ELISA and neutralization assays

CONTACTS AND LOCATIONS:
Overall Officials: Marylyn M Addo, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (2):
- Germany (2):
  - Uniklinik Köln, Cologne, North Rhine-Westphalia
  - CTC North, Hamburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grewe I, Friedrich M, Dieck ML, Spohn M, Ly ML, Krahling V, Mayer L, Mellinghoff SC, Rottstegge M, Kraemer R, Volz A, Becker S, Fathi A, Dahlke C, Weskamm LM, Addo MM. MVA-based SARS-CoV-2 vaccine candidates encoding different spike protein conformations induce distinct early transcriptional responses which may impact subsequent adaptive immunity. Front Immunol. 2024 Dec 19;15:1500615. doi: 10.3389/fimmu.2024.1500615. eCollection 2024. PMID 39749328

DOCUMENTS (1):
  • Study Protocol (2021-10-05): https://cdn.clinicaltrials.gov/large-docs/49/NCT04895449/Prot_000.pdf